CLINICAL TRIAL: NCT02069782
Title: Mother and Infant Home Visiting Program Evaluation (MIHOPE
Brief Title: Mother and Infant Home Visiting Program Evaluation
Acronym: MIHOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Collaborators: Mathematica Policy Research, Inc. (Other); Johns Hopkins University (Other); University of Georgia (Other); Columbia University (Other); James Bell Associates (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HHSP23320095644 WC
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Infant Development
Keywords: Pregnancy; postpartum programs; infant health services
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home visiting (Experimental): Home visiting programs in the United States grew from three major approaches that first became prominent in the 1960s: visits by public health nurses to promote infant and child health in disadvantaged families, Head Start home visiting to promote school readiness in hard-to-reach families, and home-based family support to promote positive parenting and prevent child abuse in high-risk families. All of these approaches sought to foster early childhood health and development by intervening in the home to support and improve socialization, health, and education practices.Today, home visiting is seen as a particularly important strategy for high-risk families who may be difficult to engage in other services.
  Interventions: Other: Home visiting

INTERVENTIONS:
Other: Home visiting — Home visits are used to assess family needs, provide support and education, and make referrals to relevant community services. The goals of the programs are to improve child health and development, promote positive parenting, prevent child maltreatment, improve maternal and child health, and increasing parental self-sufficiency.
  Other Names: HFA; PAT; EHS; NFP

SUMMARY:
MIHOPE is a multi-state study of home visiting programs authorized under the Maternal, Infant, and Early Childhood Home Visiting (MIECHV) program. The study is required by the federal Patient Protection and Affordable Care Act of 2010 (ACA), which created the MIECHV program. It is being conducted by MDRC under contract to the Administration for Children and Families within the US Department of Health and Human Services. In conducting the research, MDRC has subcontracted portions of the research to Mathematica Policy Research, Johns Hopkins University, Columbia University, University of Georgia, and James Bell Associates.

MIHOPE is randomly assigned 4,229 families nationally to home visiting services or to a comparison group that will receive referrals to other services in the community. The study is seeking to include 88 local home visiting programs (sites) that are funded through MIECHV in approximately 12 states. Data will be collected from families, local home visiting programs, and state and federal administrative data systems to assess the effects of the programs on family outcomes and to learn more about how the programs are run. Sites included in the evaluation will be using one of four national service models (Nurse Family Partnership, Healthy Families America, Parents as Teachers, and Early Head Start-Home Visiting Option) that states have chosen for most of their MIECHV funding. MIHOPE will inform the federal government about the effectiveness of the MIECHV program in its first few years of operation, and it will provide information to help states develop and strengthen home visiting programs in the future. Research findings will be disseminated through a report to Congress in 2015; reports on program impacts, implementation, and on the relationship between program features and program impacts; journal articles; and practitioner briefs.

DETAILED DESCRIPTION:
MIHOPE includes two groups of participants. First, the included 4,229 women across 88 local home visiting programs (sites) in 12 states. Women will be randomized so that half can receive home visiting services and half are in a control group that receives referrals to other services in the community. Local home visiting programs chosen for the study must meet the following criteria: (1) they have been in operation for at least two years, (2) they are receiving funds through the MIECHV program, (3) they are operating one of the four evidence-based models described earlier, and (4) there is enough need for the program's services that they can provide a control group without reducing the number of families that receive home visiting.

Families were recruited as follows. Mothers were identified as eligible for a local home visiting program by staff from that program, using the program's current procedures. If the mother appears to be eligible for MIHOPE (based on the mother's age and pregnancy status or child's age), the home visiting staff will mention that a study is going on and that someone from the study team would like to be in touch to explain the study and to see if the mother is interested in participating. The home visiting program entered the mother's address and phone number. In addition, the home visiting program provided Mathematica with the mother's name and date of birth and the child's date of birth for purposes of making sure the family is not already in the study or has not previously declined to participate in the study. The MDRC Institutional Review Board determined that a partial authorization of the HIPAA Authorization requirement was warranted for use of the mother's information for sample recruitment.

Study field staff attempted to contact the family and schedule a visit to explain the study, request their participation, and obtain informed consent for research activities. Potential study participants were asked to sign two consent forms at the beginning of the study: one to participate in the study and to allow the team to collect administrative and survey data, and a second to be video-recorded during two home visits, if assigned to the home visiting group. Mothers also provided consent to allow us to collect information from the home visiting programs about the services they receive and information from the government on various information, including Medicaid records, vital records, child welfare records, and employment and earnings information from the National Database of New Hires. If an applicant was a non-emancipated minor, assent was obtained from the minor and written consent was obtained from her parent or guardian if the parent or guardian was in the home at the time of the recruitment visit. If the parent or guardian was not in the home, verbal consent was obtained. If verbal consent was provided, the parent or guardian was mailed a copy of the assent form that the woman signed and that explains what the research entails.

After consent was provided, study staff in the family's home initiated a call to the study's survey operations center for purposes of administering a one-hour survey. The family baseline survey included information on several domains specified in the ACA: newborn health; parental health and well-being; parenting practices, attitudes, and beliefs; domestic violence; history with the criminal justice system; family economic self-sufficiency; and referral and coordination of social services. In addition, the baseline survey collected information on demographics and household composition to describe the study sample, and contact information for family members or friends who can help locate the family at follow-up if they move. The survey also contained information about the parent's expectations regarding the home visiting program, which will inform research on program implementation. While the mother was completing the baseline survey by phone, the study field staff conducted the Home Observation for Measuring the Environment (HOME) to assess the quality and amount of stimulation that the child receives in the home as well as observations of the home environment. At the end of the telephone survey, the interviewer determined whether the family was assigned to the program (home visiting program) or control group (comparison group that will receive referrals to other services in the community); the result of random assignment was sent by automated email to the point of contact at the local program.

A second round of data was collected when the child was about 15 months old. These include: (1) a one-hour telephone interview (the family follow-up survey), (2) a 30-minute video-recording of the mother and child playing with some toys (the Three Bags task), (3) a direct assessment of the child's receptive language skills (expected to take 40 minutes), (4) measurement of the child's weight and height and the mother's weight (expected to take 5 minutes), and (5) observations of the family's home environment, which will not add time to the data collection procedures. Finally, data were collected from three state systems: (1) Medicaid, (2) vital records, and (3) child welfare. Follow-up data collection plans have been approved by the federal Office of Management and Budget.

The family follow-up survey included information on several domains specified in the ACA: infant and child health; child development; parental health and well-being; parenting practices, attitudes, and beliefs; domestic violence; history with the criminal justice system; family economic self-sufficiency; and use of social services. Survey questions focused on outcomes for which previous studies of home visiting have found effects and on outcomes that would not be available from other sources (such as administrative records).

Follow-up data collection also included several types of data collected in the family's home:

1. Direct assessments of children's receptive language skills will be done using the Preschool Language Scales-5 Auditory Comprehension Scale (PLS-5), which is an individually administered test that assesses the child's ability to understand language. During the assessment, the child sat on the mother's lap while the field interviewer administered this test. At 15 months, toddlers' spoken language capabilities are only just beginning to develop. For this reason, the Auditory Comprehension subtest of the PLS-5 was used. The Auditory Comprehension cluster measures a child's ability to be attentive and respond to stimuli in the environment and to comprehend basic vocabulary or gestures.
2. During the follow-up visit, field staff used a measuring tape and a weighing scale when they conduct field visits, which they will use to obtain both the mother's weight and the child's height and weight. Direct measurements of the child's weight and length will provide information on whether the child's growth is within a normal range or exhibits early signs of unhealthy growth trajectories (i.e., risk of obesity or under-development). Measurement of the mother's weight along with self-reported height will provide information on whether the mother is obese, which is associated with a host of other health problems. When measuring weight, if the child is willing, the field interviewer will ask him or her to stand on the weighing scale by him or herself. If the child is unwilling to do so, then the staff person will obtain the mother's weight and then ask her to pick up the child and stand on the scale with the child. The mother's weight will then be subtracted from this total weight to obtain the child's weight. These measures are being collected out of concern that the mother may not accurately report her own weight and may not know her child's current weight and height.
3. The Home Observation for Measuring the Environment (HOME) - described under baseline data collection -- was conducted again at follow-up.
4. The three bags task, a direct observation of parent-child interactions, was conducted. This assessment is intended to capture the parenting constructs of parental sensitivity, cognitive stimulation, positive regard, intrusiveness, negative regard, detachment, relationship quality (degree of relatedness and mutual engagement), and boundary dissolution (parent's inability to maintain an appropriate role in his or her interaction with child). From this task, children's behaviors towards the parent will also be gathered in the context of the parent-child interaction, including engagement with the parent, sustained attention, and negativity towards the parent.

In addition, the study asked approximately 500 home visitors and 100 supervisors in the 85 sites to enroll in the study. Some supervisors may also see families and carry a caseload, acting in the capacity of both supervisor and supervisor. Program staff were identified by a local program manager and sent emails by the study team asking them to enroll in the study. Home visitors and supervisors were asked to complete a 75-minute web-based survey around the time that the site enters the study. The home visitor and supervisor baseline surveys collected information on staff characteristics and on staff perceptions of organizational factors related to service delivery; employment, supervision and program outcomes; staff beliefs about home visitor roles and responsibilities, ratings of her or his own training and skills in supervising staff to carry out activities; ratings of her or his own ability to secure supervision and professional consultation; and demographics and individual background characteristics. Individuals who are both home visitors and supervisors were asked to complete a survey that combined elements of the home visitor and supervisor surveys, and lasted about 105 minutes. Because the surveys included sensitive information, home visitors and supervisors were asked to consent to the survey and home visitors were asked to consent to videotaped interactions with families. Home visitors and supervisors were asked to provide consent through a web-based application before completing the web-based surveys.

Home visitors and supervisors were asked to complete a 75-minute web-based survey again a year after enrolling in the study. Staff who are both home visitors and supervisors were asked to complete a 105-minute web-based survey again a year after enrolling in the study. Staff follow-up surveys parallel the baseline surveys. They measured malleable respondent characteristics and perceptions of organizational factors related to service delivery.

MIHOPE has also completed two additional follow-up surveys that were conducted around the time the child turns 2 ½ and 3 ½ years old. At those two points in time, the mother - or the child's primary caregiver if the mother was not available - was asked to take part in a short survey. The survey included about 15 minutes of questions on topics such as child and parental health, parenting style, child development, and social services used. The caregiver was also asked to provide updated contact information, as well as share information about people who may know how to locate her in the future.

MIHOPE planned to conduct a kindergarten follow-up during the four school years in which children in the sample were slated to attend kindergarten: 2018-2019 (Cohort 1), 2019-2020 (Cohort 2), 2020-2021 (Cohort 3), and 2021-2022 (Cohort 4). However, due to the COVID-19 pandemic, kindergarten data collection paused during the 2020-2021 school year. It resumed during the 2021-2022 school year, when children in Cohort 3 were slated to attend first grade and children in Cohort 4 were slated to attend kindergarten. In light of the ongoing pandemic, the study team adapted the kindergarten data collection to conduct all in-home assessments virtually for Cohorts 3 and 4 during the 2021-2022 school year. To gather information on MIHOPE families' experiences during the pandemic, the study team designed and implemented a brief web survey and virtual qualitative interviews with caregivers. These data will be used to contextualize the study's kindergarten findings.

Because home visiting aims to affect a wide range of outcomes, the study team collected a wide range of data for the kindergarten follow-up, from the following data sources:

* A structured interview with the children's mothers to measure a broad set of constructs that are mostly not available from other data sources. In cases where the mother was not available (for example, because she no longer had custody of the child), data collection was conducted with the child's primary caregiver, such as the child's father. This approach was also used at the MIHOPE follow-up that occurred when children were 15 months of age.
* Direct assessments of children's language, math, and executive functioning skills conducted by trained field interviewers.
* Observations of parental warmth and children's self-regulation conducted by trained field interviewers during the direct assessment.
* Observations of mother-child interactions, such as parental sensitivity and child engagement of parent, by trained independent observers during a video-recorded semi-structured play interaction.
* A direct assessment of mothers' working memory conducted by trained field interviewers.
* A teacher survey to measure children's social and emotional development, approaches to learning, disciplinary incidents, receipt of special services, and school attendance.
* Federal administrative data on healthcare use via Medicaid.
* Federal administrative data on employment covered by the unemployment insurance system (National Directory of New Hires).
* State child welfare records.
* School records from state and local education agencies.

As mentioned previously, two additional data sources collected information about families' experiences during the COVID-19 pandemic: (1) a brief web survey was administered to families in all cohorts in September and October 2020, and (2) qualitative interviews were conducted with a subsample of 100 families who responded to the web survey between October 2020 and January 2021.

The study team will examine the effects of home visiting on 66 child and family outcomes in five outcome areas and show estimated effects for these individual outcomes in the kindergarten report. To focus the impact analyses and aid in the interpretation of the results, the study team has developed several topical research questions and will use omnibus tests to interpret the pattern of effects across the outcomes relevant to each research question. (The study team plans to use omnibus tests based on Devin Caughey, Allan Dafoe, and Jason Seawright, "Nonparametric Combination (NPC): A Framework for Testing Elaborate Theories." Journal of Politics 79, 2 2017: 688-701 to characterize patterns by accounting for the magnitude of estimated effects; they have used this approach in earlier MIHOPE analyses (see Michalopoulos et al., 2019 and Faucetta et al., 2023).) The study team will draw on the answers to these multiple topical research questions in interpreting the effects of home visiting at the kindergarten follow-up. While several topical research questions were pre-specified (shown below), additional research questions may be examined. In the kindergarten report, questions will be identified as pre-specified or not pre-specified. The research questions are listed in the section on outcomes.

MIHOPE has also begun a follow-up around the time children in the sample are in third grade, which will gather administrative data that can be used to conduct a benefit-cost analysis, impact analysis, and mediation analyses.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for home visiting program selected to be in the study
* At least 15 years old
* Pregnant or have a child under 28 weeks old

Exclusion Criteria:

* women already enrolled in home visiting (for example, with an older child)
* children in foster care in sites using EHS program model
* homeless families in sites using EHS program model
* women who speak neither English or Spanish

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4232 (Actual)
Dates: Start 2012-10; Primary Completion 2019-01 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
New pregnancy after study entry | through child's 15th month
  Mother has had one or more pregnancies since study entry
Any health encounter for injury or ingestion | through child's 15th month
  Whether the child has had an injury or ingestion that lead to a health encounter.
Number of well-child visits | through child's 15th month
  Number of well-child visits
Parental supportiveness | at child's 15th month
  Parental supportiveness measured from Three Bags interaction of parent with child
Quality of home environment | at child's 15th month
  Quality of home environment measured using the IT-HOME
Child has health insurance coverage | at child's 15th month
  Whether the child has health insurance coverage
Behavior problems | at child's 15th month
  Behavior problems total score from the BITSEA parent report
Frequency of minor physical assault of child | through child's 15th month
  Whether parent reports indicate child has been victim of minor physical assault
Frequency of psychological aggression | through the child's 15th month
  Whether parent reports indicate child has been victim of psychological aggression
Any child ED use | through child's 15th month
  Whether child has visited the ED
Language skills in the normal range | at child's 15th month
  Whether child has language skills in the normal range, as measured through a direct assessment
Parent receiving education or training | at child's 15th month
  Whether parent is receiving education or training

OTHER OUTCOMES:
New birth after study entry | When focal child is 2.5 years old and when focal child is 3.5 years old
  Mother reports having given birth to one or more children after study entry
Maternal depressive symptoms | When focal child is 2.5 years old and when focal child is 3.5 years old
  Whether mother reports depressive symptoms based on the CESD-10 scale
Health status of mother is rated "fair" or "poor" | When focal child is 2.5 years old and when focal child is 3.5 years old
  Whether mother reported her health was fair or poor
Number of child emergency department visits for accident or injury | From age 15 months to 2.5 years for the child, and from 2.5 years to 3.5 years
  Mother's report of number of visits to the ED for the child for accidents or injuries
Mother is pursuing education or training | When focal child is 2.5 years old and when focal child is 3.5 years old
  Whether the mother indicates she is currently receiving training or education
Use of yelling as a disciplinary practice | When focal child is 2.5 years old and when focal child is 3.5 years old
  Mother's report of yelling at the child as a disciplinary practice
Direct interactions between parents and home visitors | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring interactions between parents and home visitors
Children's social-emotional functioning in the home context | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring children's social-emotional functioning in the home context
Children's social-emotional functioning in school setting | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring children's social-emotional functioning in school context
Children's language, early math, and cognitive skills | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring children's cognitive skills
Parent-child interactions | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring parent-child interactions
Aggression, conflict, violence, and maltreatment | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring child maltreatment and intimate partner violence
Material hardship, employment, education, and income | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring the listed economic outcomes
Maternal mental and behavioral health | When child is in kindergarten or first grade
  Omnibus test on outcomes measuring maternal behavioral health

CONTACTS AND LOCATIONS:
Overall Officials: Charles Michalopoulos, PhD, Principal Investigator — MDRC; Virginia Knox, PhD, Principal Investigator — MDRC; Anne Duggan, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- MDRC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A restricted access file with data at baseline, 15 months, 2.5 years, and 3.5 years has been made available to researchers through ICPSR. All data were masked so that individuals cannot be identified. All data used in the study analysis were included in the file. Details about the files can be found here: https://www.icpsr.umich.edu/web/about/cms/3727.
Time Frame: Data through the 3.5 year follow-up are now available.
Access Criteria: Individuals must apply for access to the data and cannot have knowledge about any individual study participants.
URL: https://www.icpsr.umich.edu/web/about/cms/3727

REFERENCES:
- [Background] Charles Michalopoulos, Anne Duggan, Virginia Knox, Jill H. Filene, Helen Lee, Emily K. Snell, Sarah Crowne, Erika Lundquist, Phaedra S. Corso, Justin B. Ingels (2013). Revised Design for the Mother and Infant Home Visiting Program Evaluation. OPRE Report 2013-18. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Background] Charles Michalopoulos, Helen Lee, Anne Duggan, Erika Lundquist, Ada Tso, Sarah Crowne, Lori Burrell, Jennifer Somers, Jill H. Filene, and Virginia Knox. (2015). The Mother and Infant Home Visiting Program Evaluation: Early Findings on the Maternal, Infant, and Early Childhood Home Visiting Program. OPRE Report 2015-11. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Background] Charles Michalopoulos, Kristen Faucetta, Carolyn J. Hill, Ximena A. Portilla, Lori Burrell, Helen Lee, Anne Duggan, and Virginia Knox. (2019). Impacts on Family Outcomes of Evidence-Based Early Childhood Home Visiting: Results from the Mother and Infant Home Visiting Program Evaluation. OPRE Report 2019-07. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Result] Phaedra S. Corso, Justin B. Ingels, and Rebecca L. Walcott. (2022). Costs of Evidence-Based Early Childhood Home Visiting: Results from the Mother and Infant Home Visiting Evaluation. OPRE Report 2022-01. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Result] Faucetta, Kristen, Charles Michalopoulos, Ximena A. Portilla, and Kelly Saunders 2023. Checking in with Families in the Mother and Infant Home Visiting Program Evaluation. OPRE Report 2023-140. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- See also: MIHOPE Report to Congress (cited above) — https://www.mdrc.org/publication/mother-and-infant-home-visiting-program-evaluation
- See also: MIHOPE impacts at 15 months — https://www.mdrc.org/publication/impacts-family-outcomes-evidence-based-early-childhood-home-visiting
- See also: Report on costs of the intervention — https://www.mdrc.org/work/publications/costs-evidence-based-early-childhood-home-visiting
- See also: Impacts at 2.5 and 3.5 years — https://www.mdrc.org/work/publications/checking-families-mother-and-infant-home-visiting-program-evaluation
- See also: MIHOPE revised design — https://www.mdrc.org/work/publications/revised-design-mother-and-infant-home-visiting-program-evaluation